CLINICAL TRIAL: NCT02633605
Title: Comparison of First Sense Breast Exam® to the University of Toledo Mammography and Biopsy Results
Status: Completed | Type: Observational
Sponsor: First Sense Medical, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: FSM-002
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- First Sense Breast Exam
  Interventions: Device: First Sense Medical®

INTERVENTIONS:
Device: First Sense Medical®

SUMMARY:
First Sense Medical®, LLC is a medical device company developing a novel breast cancer screening tester called the First Sense Breast Exam® Tester. This radiation free tester is being developed to produce data which will be analyzed by Therma-Scan Reference Laboratory. When the tester is in production, a test will take approximately 7 minutes and will be performed in a doctor's office.

DETAILED DESCRIPTION:
This study is designed to evaluate the First Sense Breast Exam® test and the analysis by Therma-Scan. The First Sense Breast Exam® test is an adjunct to a mammogram. Currently, mammography is the standard of care in screening for breast cancer, and manual thermology is an adjunctive screening method. All of the study costs will be incurred by the sponsor and the subject will incur no costs to participate in the study. The First Sense Tester is a non-significant risk device where the tester's imaging camera makes no contact with the subjects during the entire procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female, over the age of 18 years of age.
* Asymptomatic women and women who are being screened for breast abnormality.
* Women scheduled for a mammogram or women who have had a mammogram and are given 3 days to wait in between their mammogram and scheduled biopsy and FS/TS system.
* Not pregnant or breast feeding.
* Signed Informed consent.

Exclusion Criteria:

* Subject does not meet inclusion criteria, noted above.
* Use of niacin or niacin patch.
* Use of nitroglycerin.
* Subject experienced a fever of 102°F or higher within thirty-six (36) hours of the study.
* Patients with any prior breast surgery (implants, reduction, lumpectomy, mastectomy, mastopexy, reconstruction and incisional biopsies.).
* History of breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of adult women who are having a diagnostic or screening mammogram.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

PRIMARY OUTCOMES:
Percentage of breast cancer cases detected by the new medical device (the First Sense Medical technology) | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Eleanor N. Dana Cancer Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided